CLINICAL TRIAL: NCT03321916
Title: Controlled Pilot Study for Safety and Efficacy of Subthreshold Photothermal Therapy for Patients With Macular Telangiectasia (MacTel) Type 2
Brief Title: MacTel Laser Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Lowy Medical Research Institute Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MacTelLaser1
Record Dates: First submitted 2017-10-18; First posted 2017-10-26 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Macular Telangiectasia
Keywords: MacTel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Subthreshold Photothermal Therapy (Experimental)
  Interventions: Device: 577-nm PASCAL laser
- Sham (Sham Comparator)
  Interventions: Device: 577-nm PASCAL laser

INTERVENTIONS:
Device: 577-nm PASCAL laser — The Topcon/Endpoint Management System™ is a cleared medical device commonly used in the treatment of ocular disorders.

SUMMARY:
This is a two armed Single Masked Pilot Study enrolling participants with Macular Telangiectasia Type 2 who will be randomized to undergo either a subthreshold photothermal treatment or a sham procedure to one eye. The participants will be followed for one year with visits at 1 month, 3 months, 6 months and 12 months post-treatment (laser or sham). Due to the small number of participants enrolled in this study the data will be analyzed by descriptive statistics and exploratory figures. Summary statistics will be produced for study and fellow eyes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent obtained from the participant in accordance with the local regulations;
2. Males/females 21 years of age and older but less than 80 years of age;
3. Participant must have a positive diagnosis of MacTel Type 2 in at least one eye with evidence of fluorescein leakage typical of MacTel or at least one of the other features including loss of retinal transparency/hyper-reflectivity to blue light, crystalline deposits, right angle vessels, inner/outer retinal low-reflective spaces, or hyperpigmentation not involving the center of the fovea, but no evidence of intraretinal/subretinal vascular proliferation;
4. Participant must have an Ellipsoid Zone (EZ, aka IS/OS) break in the study eye between 0.16 - 4.0 mm2 as measured on SD-OCT;
5. Participant's best-corrected visual acuity at least 55 letters (20/80) in the study eye;
6. Participant must have steady fixation in the foveal or parafoveal area of each eye, adequate pupil dilation and sufficiently clear media to perform multi-modal retinal imaging and treatment;
7. Participant must be able and willing to attend all scheduled visits.

   For Participants undergoing optional AOSLO imaging:
8. Participant should have reproducible baseline AOSLO image montages at 2 baseline imaging sessions with quality suitable to identify a minimum of 7 regions of interest (ROIs) at which reliable cone spacing measures can be made in each eye.

Exclusion Criteria:

1. Participant is unable to provide informed consent;
2. Participant is less than 21 years of age or greater than 80 years of age; (but less than 80);
3. Participant is medically unable to comply with study procedures or follow-up visits;
4. Participant received intravitreal therapy for non-neovascular MacTel in the study eye and in the fellow eye, injections no sooner than 3 months prior to study treatment;
5. Participant has nystagmus in either eye;
6. Participant has greater than 7 diopters myopia in either eye;
7. Participant has been diagnosed and treated for amblyopia in the study eye;
8. Participant has significant ocular abnormalities in either eye that prevent retinal assessment, including media opacities or cataract (up to Nuclear Sclerosis +1 is allowable);
9. Participant was a study participant in any other clinical trial of an intervention (drug or device) within the last 6 months;
10. Participant has a history of malignancy that would compromise the 12 month study survival; or
11. Participant has, in the opinion of the Investigator, any physical or mental condition that would increase the patient's risk of participation in the study or may interfere with the study procedures, evaluations and outcome assessments;
12. Presence of signs of advanced retinal/vascular disease in the study eye, such as CNV, haemorrhages or macular atrophy based on OCT or FAF;
13. Previous macular laser treatment in either eye;
14. Any previous ocular condition that may be associated with a risk of developing macular oedema;
15. Vitreomacular traction determined clinically and/or by OCT, which in the opinion of the investigator contributes to the macular oedema (associated or causing a detachment of the fovea) in the study eye;
16. Presence of other macular disease such as epiretinal membrane in the study eye;
17. Ocular or periocular infections;
18. Planned intra-ocular surgery in the study eye within one year; and
19. Patient is unavailable for follow-up visits.

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 months post treatment
  To evaluate the safety and tolerability of subthreshold photothermal therapy in patients with MacTel Type 2 as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Change from baseline cone density as measured by confocal adaptive optics (AOSLO) | 1 year
  To evaluate the biological activity of subthreshold photothermal therapy in patients with MacTel Type 2.
Change in size of ellipsoid zone break area as measured by spectral domain optical coherence tomography (SD-OCT) | 1 year
  To evaluate the biological activity of subthreshold photothermal therapy in patients with MacTel Type 2.
Development or extension post therapy of areas of deficiency in cones as measured by AOSLO | 1 year
  To evaluate the biological activity of subthreshold photothermal therapy in patients with MacTel Type 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin & Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes